CLINICAL TRIAL: NCT01481532
Title: Open Label Phase I Clinical Trial of Crotoxin in Patients With Advanced Cancer Using an Intravenous Route of Administration
Brief Title: Open Label Clinical Trial of Intravenous Crotoxin Part 3
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Celtic Biotech Ltd (Industry)
Collaborators: Institut de Cancérologie de l'Ouest (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRTX01
Record Dates: First submitted 2011-10-11; First posted 2011-11-29 (Estimated); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Cancer
Keywords: Antineoplastic agent
MeSH Terms: conditions — Neoplasms | interventions — Crotoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cohort 3 (Experimental): The third cohort will include up to 24 patients with Crotoxin doses of 0.2 to 1.32 mg per m2 in which the dose escalation speed will be faster. Drug is administered over 3 + 4 day intervals using ambulatory infusion pumps; treating on an outpatient basis. Subjects will receive increasing doses over the course of 28 treatment days (8 dose levels). Dose escalation will continue if DLT is not established
  Interventions: Drug: Crotoxin

INTERVENTIONS:
Drug: Crotoxin — Intra patient dose escalation
  Other Names: CB-24

SUMMARY:
The primary objective of the study is to assess whether human subjects can be made tolerant to intravenously administered Crotoxin and achieve higher and more therapeutically effective doses levels without the previously reported adverse effects associated with bolus i.m. administration.

DETAILED DESCRIPTION:
Crotoxin has been shown to induce neurotoxic tolerance in animals allowing them to receive high doses associated with effective anti-tumor activity in the absence of adverse side effects.

The study plans to demonstrate this effect in human subjects using two dose escalation protocols; slow and fast. It is believed that this approach will prevent toxic side effects to subjects.

The route of administration has not been employed clinically and is designed to avoid the myonecrotic effects of intramuscular injections. The target maximum dose is almost five times that of the previously reported MTD.

The revised protocol incorporates continuous infusion with a mobile pump and includes active suppression of the allergic reaction by pre-treatment administration of antihistamines.

ELIGIBILITY:
Subjects will:

1. Be adult patients with histologically confirmed advanced solid tumors (excluding basal cell, colon, pancreatic and stomach cancers) who have progressed despite standard therapy, or for whom no standard therapy exists.
2. Have an ambulatory PS (ECOG 0-1).
3. Have tumor evaluation made within 28 days before study drug administration
4. Have completed radiotherapy or chemotherapy or any other anticancer therapy (including experimental therapy) more than 4 weeks prior to enrolment into the trial and must have recovered from all acute side effects of these treatments
5. Have a life expectancy greater than 3 months
6. Have an age ≥ 18 years
7. Have normal marrow function with the following haematological parameters normal; Hb ≥10g/dl, WBC ≥4.0 x10E9/L, neutrophil count ≥ 2.0 x 10E9/L and platelets ≥100 x10E9 /L
8. Have no medically significant impairment of cardiac or respiratory functions<
9. Have adequate hepatic function with Total bilirubin 1.5 x N and Transaminases < 2.5 x N (< 5 x N in case of liver metastasis).
10. Have no history of prior severe allergic reactions to venoms
11. Have Creatinine clearance > 50 mL/min.
12. Be on stable doses of any drugs which may affect hepatic drug metabolism or renal drug excretion (e.g.--non-steroidal anti-inflammatory drugs, barbiturates, narcotic analgesics, probenecid). Such drugs should not be initiated while the patient is participating in this study.
13. Not be pregnant or planning to become pregnant
14. Not known to have brain metastases or leptomeningeal involvement. CT-scan or MRI is not required to rule this out unless there is clinical suspicion of central nervous system involvement
15. Not have pleural effusion/ ascites, cystic lesions or bone metastases, as the only assessable lesions
16. Not have a history of other malignancies, except for patients with a cancer free interval of > 5 years after treatment completion, patients with prior history of adequately treated basal cell carcinoma of the skin or carcinoma in situ of the cervix
17. Not have had recent major surgery (within 21 days).
18. Not have a recent history of weight loss > 10% of current body weight.
19. Not have serious intermittent medical illnesses which would interfere with the ability of the patient to carry out the treatment program.
20. Not be on chronic steroid medication (> 20mg/day)
21. Not have primary or paraneoplastic myasthenia gravis
22. Be free of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule;
23. Will agree to participate in the study prior to starting with any specific study procedure, after having signed written informed consent.
24. Be patients of childbearing age willing to use contraceptive for the duration of the study
25. Not live alone and live no further than approximately 30 km away from the hospital, and for the study duration have continuous access to the use of mobile telephone in case of medical emergency

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Tolerability of intra-patient dose escalation | 28 days
  Assess the safety and tolerability of Crotoxin administered intravenously to Stage IV cancer patients using intra-patient dose escalation procedure.
Confirmation of the induction of drug tolerance | 28 days
  Confirm in a controlled phase I trial that human subjects can be made tolerant to intravenously administered Crotoxin thereby reducing the potential for adverse drug effects

SECONDARY OUTCOMES:
Assessment of drug efficacy | 112 days
  Document any objective anti-tumour responses that occur in patients treated on this protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Campone, MD, Ph.D, Principal Investigator — INSTITUT DE CANCEROLOGIE DE L'QUEST, Saint Herblain, France
Locations (1):
- Institut de Cancérologie de l'Ouest, Saint-Herblain, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Medioni J, Brizard M, Elaidi R, Reid PF, Benlhassan K, Bray D. Innovative design for a phase 1 trial with intra-patient dose escalation: The Crotoxin study. Contemp Clin Trials Commun. 2017 Jul 23;7:186-188. doi: 10.1016/j.conctc.2017.07.008. eCollection 2017 Sep. PMID 29696184
- [Background] Gil-Delgado M, Paul G, Bray DH, Delgado F, Spano JP, Idbaih A, Reid PF, Benlhassan K, Diaw C, Khayat D. Continuous i.v. Crotoxin in advanced cancer: Intra-patient dose escalation. Cancer Res (2018) 78 (13_Supplement): CT071.